CLINICAL TRIAL: NCT00000823
Title: A Multicenter Phase II Double-Blind Exploratory Study to Evaluate Differences Among Various Zidovudine/Didanosine Regimens on Quantitative Measures of Viral Burden in Relatively Early HIV-1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 276; 11252 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Zidovudine; Drug Administration Schedule
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To determine the relative antiviral activity and safety of zidovudine ( AZT ) and didanosine ( ddI ) alone and in combination, as well as in various sequences of administration.

The relative efficacy of the approved antiretrovirals in early HIV-1 disease is unclear; thus, a study is needed to evaluate the ability of these various nucleoside analogs to limit pathogenicity.

DETAILED DESCRIPTION:
The relative efficacy of the approved antiretrovirals in early HIV-1 disease is unclear; thus, a study is needed to evaluate the ability of these various nucleoside analogs to limit pathogenicity.

Patients undergo observation for 2 weeks, then are randomized to one of six treatment arms to receive ddI alone or in sequence or combination with AZT for 16-32 weeks, followed by 4 weeks of post-treatment evaluation. The regimens are: ddI alone for 32 weeks; AZT for 16 weeks followed by ddI for 16 weeks; AZT for 16 weeks followed by AZT/ddI combination for 16 weeks; ddI for 16 weeks followed by AZT for 16 weeks; AZT/ddI combination for 32 weeks; and placebo for 32 weeks.

PER AMENDMENT 6/18/96: NOTE: Patients enrolled under version 3 of the study will terminate treatment at week 16 and have a 4 week follow up.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositivity.
* CD4 count >= 550 cells/mm3.
* Asymptomatic disease.
* No prior antiretroviral therapy.
* Consent of parent or guardian if less than 18 years old.

PER AMENDMENT 6/18/96:

* Patients with an undocumented history of oral candidiasis or a history of candidiasis that was antibiotic associated may enroll.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Medical condition that precludes study compliance.

Concurrent Medication:

Excluded:

* Antiretrovirals other than study drugs.
* Biologic response modifiers including erythropoietin and G-CSF.
* Systemic corticosteroids.
* Systemic cytotoxic chemotherapy.
* Intravenous pentamidine.

Concurrent Treatment:

Excluded:

* Systemic radiation therapy.

Patients with the following prior conditions are excluded:

* History of grade 2 or worse peripheral neuropathy.
* History of pancreatitis or factors predisposing to pancreatitis.

Prior Medication:

Excluded:

* Prior antiretrovirals.
* Systemic immunomodulators (e.g., gp120, gp160, IL-2, interferons) within 3 months prior to study entry.

Chronic alcoholism.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85
Dates: Study Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Collier AC, Study Chair; Johnson V, Study Chair
Locations (22):
- United States (22):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Illinois Masonic Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Washington, Seattle, Washington